CLINICAL TRIAL: NCT00884052
Title: Pharmacokinetic and Safety Trial of Intravenous Levetiracetam in the Treatment of Neonatal Seizures
Acronym: Keppra
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Richard H. Haas (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor-Investigator, Richard H. Haas, Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Thrasher 02825-1; NCT00461409 (obsolete NCT alias)
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2020-03-26 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Seizures; Disorder of Fetus or Newborn
Keywords: Neonatal seizures
MeSH Terms: conditions — Seizures; Fetal Diseases | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- levetiracetam dose escalation (Experimental): 6 Babies in Phase 1-Received Dose 1: 20 mg/kg; 5 mg/kg daily 12 Babies in Phase 2-Received Dose 2: 40 mg/kg; 10 mg/kg/day
  Interventions: Drug: Low dose levetiracetam; Drug: High dose levetiracetam

INTERVENTIONS:
Drug: Low dose levetiracetam — 20 mg/kg loading dose; 5 mg/kg daily for 7 days.
  Other Names: Keppra
Drug: High dose levetiracetam — 40 mg/kg IV load; 10 mg/kg/day maintenance
  Other Names: Keppra

SUMMARY:
The hypothesis is that a loading dose of 20 mg/kg and a maintenance dose of 5 mg/kg of Levetiracetam is going to be safe and effective in the treatment of seizures in neonates.

DETAILED DESCRIPTION:
In adults, drug clearance is less than half of the glomerular filtration rate and the drug half-life is 6-8 hours. Renal function in infants at birth is characterized by immature glomerular filtration and is only 20% that of older children. The specific esterase responsible for levetiracetam hydrolysis has not been identified and its expression in newborn infants is unknown. Depending on its activity, the expected infant total levetiracetam clearance will likely be between 15-45% of older populations. However, due to immaturity in levetiracetam clearance in infants, accumulation with multiple dosing is possible. Therefore the maintenance dose is reduced compared to older children according to the anticipated impaired clearance.

These anticipated differences in levetiracetam clearance and volume of distribution, will likely result in a prolonged drug half-life of 10-30 hours in infants. This prolonged elimination will require longer sampling to adequately characterize levetiracetam pharmacodynamics in this population.

The primary intent of the data analysis is to determine levetiracetam pharmacokinetics in newborn infants and predict the dosage necessary to maintain concentrations similar to those seen with effective therapy in other populations. Graphs of serum concentration vs. time will be plotted for levetiracetam for each infant. Mean serum drug concentration vs. time curves will also be constructed. Summary statistics (i.e., n, mean, standard deviation, minimum, maximum, and coefficient of variation) will be calculated for serum concentrations for each time point and each dose level.

ELIGIBILITY:
Inclusion Criteria:

* Newborns admitted to the UCSD, Children's Hospital or Sharp Mary Birch NICUs with seizures.
* Term infants (gestational age greater than or equal to 37 weeks.
* > 2500 grams (max blood for study 6mL =3%).
* Postnatal age 14 days or less.
* Serum creatinine less than 1.2 at time of enrollment.
* Received loading dose of phenobarbital 20mg/kg.
* Are still experiencing either clinical or electroencephalographic seizures despite this therapy.
* For whom parental consent to participate in the study is obtained.

Exclusion Criteria:

* Biochemical abnormality - hypoglycemia, hypocalcemia-that when treated result in seizure cessation.
* Severe hypoxic ischemic injury likely to result in imminent death
* The only significant exclusions that will be made in recruitment and enrollment will be the exclusion of infants who are judged by the attending neonatologist to be so critically ill that death is imminent and benefit from neonatal intensive care is very unlikely.
* No rule-based criteria, (using lab or clinical parameters) adequately capture the complete nature of this clinical assessment.
* In general any child receiving active treatment with head cooling will not be excluded.
* Mechanical ventilation and/or the use of inotropic agents to support blood pressure will not be exclusion criteria.

Ages: 1 Minute to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2007-04; Primary Completion 2011-03 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Haas, MD, Principal Investigator — University of Calfornia, San Diego
Locations (1):
- University of California, San Diego Medical Center / Neonatal Intensive Care Unit (NICU), San Diego, California, United States

REFERENCES:
- [Result] Sharpe CM, Capparelli EV, Mower A, Farrell MJ, Soldin SJ, Haas RH. A seven-day study of the pharmacokinetics of intravenous levetiracetam in neonates: marked changes in pharmacokinetics occur during the first week of life. Pediatr Res. 2012 Jul;72(1):43-9. doi: 10.1038/pr.2012.51. Epub 2012 Apr 11. PMID 22495532

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment over 2 years from neonatal intensive care units
Groups:
- Levetiracetam Low Dose: Levetiracetam 20 mg/kg load followed by 5 mg/kg/day for 7 days. n=6
- Levetiracetam High Dose: Levetiracetam 40 mg/kg load followed by 10 mg/kg/day for 7 days. n=12
Period: Overall Study
Arm/Group | Levetiracetam Low Dose | Levetiracetam High Dose
Started | 6 | 12
Completed | 6 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Neonates 14 days old or less. Newborns with Seizures Despite Phenobarbital Treatment.
Groups:
- Levetiracetam Dose Escalation: Escalation of dose after 6 patients treated to 40 mg/kg IV load and 10mg/kg/day maintenance
  levetiracetam : 20 mg/kg loading dose; 5 mg/kg daily for 7 days.
  levetiracetam : 40 mg/kg IV load; 10 mg/kg/day maintenance
Arm/Group | Levetiracetam Dose Escalation
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 18
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Days] | 2.44 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 13
  New Zealand | 5

OUTCOME MEASURES:

1. Primary Outcome: Drug Clearance
Time Frame: Day 1 and Day 7
Population: Subjects were grouped together to improve the reliability of the analysis. The publication of these results reported a grouped analysis because of the small number of subjects in the low dose group, The groups were not analyzed individually.
Measure: Mean (Standard Deviation); unit: ml/min/kg
Groups:
- All Participants: Participants in both low dose and high dose arms are reported together
Arm/Group | All Participants
Number analyzed (Participants) | 18
ml/min/kg
  Day 1 | 0.71 (0.27)
  Day 7 | 1.31 (0.35)

2. Secondary Outcome: Levetiracetam Treated Number of Participants With Serious Adverse Events
Time Frame: 7 Days
Measure: Count of Participants; unit: Participants
Groups:
- Levetiracetam Low Dose: 6 Babies in Phase 1-Received Dose 1: 20 mg/kg; 5 mg/kg daily
  levetiracetam: 20 mg/kg loading dose; 5 mg/kg daily for 7 days.
- Levetiracetam High Dose: 12 Babies in Phase 2-Received Dose 2: 40 mg/kg; 10 mg/kg/day
Arm/Group | Levetiracetam Low Dose | Levetiracetam High Dose
Number analyzed (Participants) | 6 | 12
Participants | 0 | 1

3. Primary Outcome: Drug Half Life
Time Frame: Day 1 and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | All Participants
Number analyzed (Participants) | 18
hr
  Day 1 | 18.5 (7.1)
  Day 7 | 9.1 (2.0)

ADVERSE EVENTS:
Time Frame: 7 days
Description: Mild adverse events which resolved spontaneously and were possibly related to treatment with LEV included mild sedation in 2 subjects, feeding difficulty in 3 subjects, mild apnea and bradycardia in one subject and decreased urine output responding to furosemide in one subject. In no case was LEV thought causative of an adverse event.
Groups:
- All Participants: There were two arms (1) Levetiracetam 20 mg/kg load followed by 5 mg/kg/day for 7 days. n=6 and (2) Levetiracetam 40 mg/kg load followed by 10 mg/kg/day for 7 days. n=12, however the data collected regarding adverse events was not recorded according to group, so all participants are reported together.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 7/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=18)
Respiratory failure (Nervous system disorders) | 1 (1) — A baby with a CNS developmental anomaly on high dose phenobarbital also treated with levetiracetam for seizures required intubation and ventilation for respiratory failure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=18)
Sedation (Nervous system disorders) | 2 (2) — Mild adverse events which resolved spontaneously and were possibly related to treatment with LEV included mild sedation in 2 subjects. In no case was LEV thought causative of an adverse event.
Feeding Difficulty (General disorders) | 3 (3) — Mild adverse events which resolved spontaneously and were possibly related to treatment with LEV included feeding difficulty in 3 subjects. In no case was LEV thought causative of an adverse event.
Apnea and Bradycardia (Nervous system disorders) | 1 (1) — Mild adverse events which resolved spontaneously and were possibly related to treatment with LEV included mild apnea and bradycardia in one subject . In no case was LEV thought causative of an adverse event.
Decreased Urine output (Renal and urinary disorders) | 1 (1) — Mild adverse events which resolved spontaneously and were possibly related to treatment with LEV included and decreased urine output responding to furosemide in one subject. In no case was LEV thought causative of an adverse event.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No